CLINICAL TRIAL: NCT06313931
Title: Effects of Cognitive-motor Training on Cognition, Depression and Daily Functioning in Patients With Mild Cognitive Impairment (MCI): A Randomized Controlled Trial
Brief Title: Effects of Cognitive-motor Training on Cognition, Depression and Daily Functioning in Patients With Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Guillermo Palacios, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTI-IIDI-074-2023
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Immersive Virtual Reality; Instrumental Activities of Daily Living; Motor-cognitive Training; Geriatric Depression
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group
  Interventions: Device: cognitive training via immersive virtual reality; Other: motor stimulation
- Control group (Active Comparator): Control group
  Interventions: Other: cognitive training via paper and pencil; Other: motor stimulation

INTERVENTIONS:
Device: cognitive training via immersive virtual reality — 20 minutes per session, twice a week for six weeks (totaling 12 sessions), using the cupboard task application.
  Arms: Experimental group
Other: cognitive training via paper and pencil — 20 minutes per session, twice a week for six weeks (totaling 12 sessions), using cards.
  Arms: Control group
Other: motor stimulation — motor stimulation for 12 sessions (20 minutes per session)

SUMMARY:
This randomized controlled trial evaluated the effectiveness of an immersive virtual reality (IVR) application (focused on a daily activity) to train cognitive functions and its impact on depression and the ability to perform activities of daily living (ADL) in patients with mild cognitive impairment (MCI). With a dose of two sessions per week during six weeks, the study showed significant improvements in cognitive functions and reduction in depression, with notable effects in the experimental group. This underscores the potential of IVR as a valuable tool in the management of MCI.

DETAILED DESCRIPTION:
Background:

The increase in cases of MCI underlines the urgency of finding effective methods to slow its progression. Given the limited effectiveness of current pharmacological options to prevent or treat the early stages of this deterioration, non-pharmacological alternatives are especially relevant.

Aim: The study aimed to evaluate the effectiveness of an immersive virtual reality (IVR) application, focused on an activity of daily living (ADL), to train cognitive functions and its impact on depression and the ability to perform ADL in patients with MCI. IVR is presented as an innovative tool with the potential to offer a promising non-pharmacological approach.

Methods:The researchers implemented a 40-minute-long intervention, twice a week for six weeks (totaling 12 sessions), using the cupboard task (based on IVR). The study included the participation of individuals with MCI, randomly distributed into control (n=12) and experimental (n=14) groups. The majority in the control group were women (75%), with a mean age of 77.67 years, and in the experimental group, women represented 57.14%, with a mean age of 74.86 years. Cognitive functions, depression, and the ability to perform ADLs were assessed. The scales used were: the Spanish version of the Montreal Cognitive Assessment (MoCA-S), the Short Geriatric Depression Scale (SGDS-S) and the Instrumental Activities of Daily Living Scale. (IADL-S), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Community-dwelling, not in nursing homes
* Physically functional
* Understanding and voluntary consent
* Mild Cognitive Impairment (MCI)
* MoCA score of 19-25

Exclusion Criteria:

* Clinical dementia diagnosis
* MoCA ≤ 18 indicating probable dementia
* Neurological disorders including stroke or TBI in the last year
* History of mental/psychiatric disorders
* Substance abuse
* Difficulty using VR headset and controllers
* Medical conditions affecting trial participation
* Visual/hearing impairments
* Communication difficulties

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Spanish version of the Montreal Cognitive Assessment (MoCA-S) | 6 weeks
  Scores in the MoCA-S scale. Higher scores mean a better outcome.
Short Geriatric Depression Scale (SGDS-S) | 6 weeks
  Scores in the SGDS scale. Higher scores mean a worse outcome.
Instrumental Activities of Daily Living Scale (IADL-S) | 6 weeks
  Scores in the IADL scale. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Palacios, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Teruel, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buele J, Aviles-Castillo F, Del-Valle-Soto C, Varela-Aldas J, Palacios-Navarro G. Effects of a dual intervention (motor and virtual reality-based cognitive) on cognition in patients with mild cognitive impairment: a single-blind, randomized controlled trial. J Neuroeng Rehabil. 2024 Aug 1;21(1):130. doi: 10.1186/s12984-024-01422-w. PMID 39090664